CLINICAL TRIAL: NCT07349537
Title: Phase 1/1b, Multicenter, Open-Label, Study of RMC-5127 in Patients With Advanced KRAS G12V-Mutant Solid Tumors
Brief Title: Study of RMC-5127 in Patients With Advanced KRAS G12V-Mutant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-5127-001
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Pancreatic Adenocarcinoma; Pancreatic Ductal Adenocarcinoma (PDAC); PDAC; CRC; NSCLC; Pancreatic Cancer; Lung Cancer (NSCLC); Advanced Solid Tumors
Keywords: Advanced Solid Tumors; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; PDAC; Colorectal Cancer; CRC; Lung Cancer; Non-small Cell Lung Cancer; NSCLC; RAS; KRAS; RAS Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Lung Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: RMC-5127 Monotherapy (Experimental): Dose Escalation and Dose Expansion
  Interventions: Drug: RMC-5127
- Arm B: RMC-5127 + Daraxonrasib Combination (Experimental): Dose Escalation and Dose Expansion
  Interventions: Drug: RMC-5127; Drug: daraxonrasib
- Arm C: RMC-5127 + Cetuximab Combination (Experimental): Dose Escalation and Dose Expansion
  Interventions: Drug: RMC-5127; Drug: cetuximab

INTERVENTIONS:
Drug: RMC-5127 — oral tablets
Drug: daraxonrasib — oral tablets
  Arms: Arm B: RMC-5127 + Daraxonrasib Combination
Drug: cetuximab — IV infusion
  Arms: Arm C: RMC-5127 + Cetuximab Combination

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of RMC-5127 as a monotherapy and in combination with either daraxonrasib or cetuximab in adults with KRAS G12V-mutant solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/1b study of RMC-5127 in adults with advanced KRAS G12V-mutant solid tumors to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary clinical activity. The study consists of three arms: RMC-5127 monotherapy arm, RMC-5127 plus daraxonrasib combination arm, and RMC-5127 plus cetuximab combination arm. All arms consist of two parts: Part 1- dose exploration and Part 2- dose expansion. Both parts of the monotherapy arm may include Food Effect Cohorts.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and has provided informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Pathologically documented, locally advanced or metastatic KRAS G12V-mutated solid tumor malignancy.
* Received and progressed or been intolerant to prior standard therapy (including targeted therapy) appropriate for tumor type and stage.
* Measurable per RECIST v1.1
* Adequate organ function (bone marrow, liver, kidney, coagulation).
* Able to take oral medications.

Exclusion Criteria:

* Primary central nervous system (CNS) tumors
* Prior therapy with KRAS G12V inhibitor or direct RAS-targeted therapy (eg. degraders and/or inhibitors).
* Any conditions that may affect the ability to take or absorb study drug.
* Major surgery within 28 days prior to receiving study drug(s).
* Patient is unable or unwilling to comply with protocol-required study visits or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) | Up to approximately 3 years
  Number of patients with AEs as assessed by Common Terminology Criteria for Adverse Events CTCAE v5
Changes in vital signs | Up to approximately 3 years
  Number of patients with changes from baseline in vital signs
Changes in electrocardiogram (ECG) test values | Up to approximately 3 years
  Number of patients with changes from baseline in ECG test values
Changes in clinical laboratory test values | Up to approximately 3 years
  Number of patients with changes from baseline in clinical laboratory test values
Dose Limiting Toxicities | Up to 28 days
  Number of patients with dose limiting toxicities

SECONDARY OUTCOMES:
Cmax concentrations of RMC-5127 and daraxonrasib | Up to Cycle 5 Day 1 (each cycle is up to 28 days)
  Maximum blood concentration (Cmax) of RMC-5127 as monotherapy and in combination with daraxonrasib or cetuximab, and Cmax of daraxonrasib in combination with RMC-5127 over time as applicable
Tmax concentration of RMC-5127 and daraxonrasib | Up to Cycle 5 Day 1 (each cycle is up to 28 days)
  Time to reach maximum blood concentration (Tmax) of RMC-5127 as monotherapy and in combination with daraxonrasib or cetuximab, and Tmax of daraxonrasib in combination with RMC-5127 over time as applicable
AUC concentrations of RMC-5127 and daraxonrasib | Up to Cycle 5 Day 1 (each cycle is up to 28 days)
  Area under the blood concentration time curve (AUC) of RMC-5127 as monotherapy and in combination with daraxonrasib or cetuximab, and AUC of daraxonrasib in combination with RMC-5127 over time as applicable
Ratio of accumulation of RMC-5127 | Up to Cycle 5 Day 1 (each cycle is up to 28 days)
  Ratio of accumulation of RMC-5127 from a single dose to steady state with repeated dosing as monotherapy and in combination with darabxrasib or cetuximab over time as applicable
Half-Life of RMC-5127 and daraxonrasib | Up to Cycle 5 Day 1 (each cycle is up to 28 days)
  Elimination Half-Life (t1/2) of RMC-5127 as monotherapy and in combination with daraxonrasib or cetuximab, and t1/2 of daraxonrasib in combination with RMC-5127 over time as applicable
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR per response evaluation criteria in solid tumors (RECIST) v1.1
Duration of Response (DOR) | Up to approximately 3 years
  DOR per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - START Midwest, Grand Rapids, Michigan
  - NEXT - Dallas, Dallas, Texas
  - NEXT, San Antonio, Texas
  - START - San Antonio, San Antonio, Texas
  - NEXT - Virginia, Fairfax, Virginia